CLINICAL TRIAL: NCT04941703
Title: Investigation of Choice Alteration of the Gut Metagenome on COVID-19 Severity
Brief Title: "CHANGE COVID-19 Severity"
Acronym: CHANGE
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Recruitment issues after COVID-19 abated; not enough hypoxic patients to meet criteria.
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Wonder Drake, Wonder Drake, MD, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 210598
Record Dates: First submitted 2021-06-24; First posted 2021-06-28 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: COVID-19 Infection
MeSH Terms: conditions — COVID-19 | interventions — magnesium citrate; Probiotics

STUDY DESIGN:
Intervention Model Description: Blinded, single-center, placebo-controlled randomized clinical trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Magnesium Citrate plus a Probiotic Arm: (Experimental): Participants assigned to the magnesium citrate plus a probiotic arm will receive 1 bottle of magnesium citrate 296 mL PO once to be taken within a 4-hour period, (about 10 oz.). Because magnesium citrate remains within the intestinal lumen, a second bottle can be provided if there is limited bowel movement. Patients will be asked to take 2 capsules of probiotics twice daily for six days or until discharge, whichever is earlier.
  Interventions: Drug: Magnesium Citrate plus probiotic
- Placebo (Placebo Comparator): Participants randomized to the placebo arm will receive matching placebo 296 mL PO once to be taken within a 4-hour period, (about 10 oz.) and 2 cellulose capsules twice daily for six days or until discharge, whichever is earlier. The placebo will be flavored to match the taste of the interventional arm.
  Interventions: Drug: Magnesium Citrate plus probiotic

INTERVENTIONS:
Drug: Magnesium Citrate plus probiotic — 296 ml magnesium citrate

SUMMARY:
We are conducting an investigator-initiated, single center, blinded, placebo-controlled, randomized clinical trial evaluating magnesium citrate combined with a probiotic for the treatment of adults hospitalized with COVID-19.

DETAILED DESCRIPTION:
We are conducting an investigator-initiated, single center, blinded, placebo-controlled, randomized clinical trial evaluating magnesium citrate combined with a probiotic for the treatment of adults hospitalized with COVID-19. Patients, treating clinicians, and study personnel will all be blinded to study group assignment.

This research study is being done to determine if taking oral magnesium citrate and a probiotic will improve the outcome of adults hospitalized with COVID-19. In this study, half of the participants will receive magnesium citrate plus a probiotic and half will receive a placebo randomized 1:1. You will be placed in one of these 2 groups randomly, like the flip of a coin. The investigational arm will receive one 10 oz. bottle of magnesium citrate to drink once and 2 oral probiotic capsules to be taken twice a day for 6 days. We will also collect a blood sample on Day 1 and Day 7 for CD4+ and CD8+ evaluation and will be collecting data on each participants COVID-19 infection progression during hospitalization.

Assessments for this study will be done on day 7 and day 29 if the participant is still hospitalized at those time points. If they have been discharged from the hospital before these assessments, we will do these by phone. Each participant will also be contacted at 3 months to assess how they are doing. There will be no compensation for taking part in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Currently hospitalized or in an emergency department with anticipated hospitalization.
3. Symptoms of acute respiratory infection, defined as one or more of the following:

   1. Cough
   2. Fever (> 37.5° C / 99.5° F)
   3. Shortness of breath (operationalized as any of the following: subjective shortness of breath reported by patient or surrogate; tachypnea with respiratory rate ≥22 /minute; hypoxemia, defined as SpO2 <92% on room air, new receipt of supplemental oxygen to maintain SpO2 ≥92%, or increased supplemental oxygen to maintain SpO2 ≥92% for a patient on chronic oxygen therapy).
   4. Sore throat
   5. Anosmia
4. Laboratory-confirmed SARS (Severe acute respiratory syndrome-Coronavirus 2 (SARS CoV-2) infection within 10 days prior to randomization
5. Ability to manage own stool care

Exclusion Criteria:

1. Prisoner
2. Pregnancy
3. Breast feeding
4. Current infectious or noninfectious diarrheal illness
5. Unable to randomize within 21 days after onset of acute respiratory infection symptoms
6. Unable to randomize after hospital arrival
7. Colonic obstruction
8. Unresolved hypovolemia
9. CrCl <30ml/min
10. Hypermagnesemia
11. Diagnosis of Long QT syndrome
12. Known allergy to magnesium citrate or probiotic
13. Unresolved electrolyte imbalance such as hypokalemia or hypocalcemia. The patient can be enrolled if electrolytes are corrected and sustained.
14. Receipt of >1 dose of magnesium citrate or any other colonic cleanser in the 7 days prior to enrollment
15. Inability to receive enteral medications
16. Refusal or inability to be contacted on Day 15 for clinical outcome assessment if discharged prior to Day 15
17. Concurrent medical illness that interferes with clinical assessment Previous enrollment in this trial
18. The treating clinical team does not believe equipoise exists regarding the use of magnesium citrate plus a probiotic for the treatment of this patient.
19. Participating in any other COVID-19 therapeutic trial
20. Allergic to soy.
21. Lactose intolerant.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2022-06-25 (Actual); Study Completion 2022-06-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Magnesium Citrate Plus a Probiotic Arm: | Placebo
Started | 8 | 10
Completed | 8 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: In additional to reporting data for the full trial population we will also report data separately for patients randomized in the ICU (who tend to be more severely ill) and those randomized outside the ICU (who tend to be less severely ill) as well as those with duration of symptoms ≤5 days prior to randomization and those with >5 days of symptoms prior to randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Magnesium Citrate Plus a Probiotic Arm: | Placebo | Total
Number analyzed (Participants) | 8 | 10 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 9 | 16
  >=65 years | 1 | 1 | 2
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 67.5 [62.8 to 69.6] | 62.0 [48.3 to 72.5] | 66.0 [56.0 to 70.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 7 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 7 | 8 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 7 | 6 | 13
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: COVID Ordinal Outcome Scale
Description: Outcome measured clinical status of the participant defined by the COVID Ordinal Outcome Scale on Day 7:
  0 = Uninfected, no viral RNA detected
  1. = Asymptomatic, viral RNA detected
  2. = Symptomatic, independent
  3. = Symptomatic, assistance needed
  4. = Hospitalized, no oxygen needed
  5. = Hospitalized, oxygen by mask or nasal prongs
  6. = Hospitalized, oxygen by NIV or high flow
  7. = Intubation and mechanical ventilation, pO2/FiO2 ≥150 or SpO2/FiO2 ≥200
  8. = Mechanical ventilation, pO2/FiO2 <150 (SpO2/FiO2 <200) or vasopressors
  9. = Mechanical ventilation, pO2/FiO2 <150 and vasopressors, dialysis or ECMO
  10. = Dead
Time Frame: Baseline through Day 7 after completion of therapy
Population: 2 Participants in the Magnesium Citrate arm and 3 participants in the placebo arm were discharged prior to Day 7. No data was collected from them for this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Magnesium Citrate Plus a Probiotic Arm: | Placebo
Number analyzed (Participants) | 6 | 7
Participants
  Outcome Score = 0 | 0 | 0
  Outcome Score = 1 | 0 | 0
  Outcome Score = 2 | 1 | 1
  Outcome Score = 3 | 2 | 1
  Outcome Score = 4 | 0 | 0
  Outcome Score = 5 | 1 | 1
  Outcome Score = 6 | 2 | 4
  Outcome Score = 7 | 0 | 0
  Outcome Score = 8 | 0 | 0
  Outcome Score = 9 | 0 | 0
  Outcome Score = 10 | 0 | 0

2. Secondary Outcome: Change in Oxygen Requirements From Baseline to Day 7 by Treatment Group
Description: Measured by liters of oxygen per minute to maintain saturation above 90%
Time Frame: baseline and 7 days
Measure: Median (Inter-Quartile Range); unit: liters per minute
Arm/Group | Magnesium Citrate Plus a Probiotic Arm: | Placebo
Number analyzed (Participants) | 6 | 7
liters per minute | 2.00 [0 to 6] | 9.00 [5.00 to 15.00]

ADVERSE EVENTS:
Time Frame: The Investigators will determine daily if any adverse events occur during the period from enrollment through study day 7 or hospital discharge, whichever occurs first.
Arm/Group | Magnesium Citrate Plus a Probiotic Arm: | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 0/8 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-13): https://cdn.clinicaltrials.gov/large-docs/03/NCT04941703/Prot_SAP_001.pdf
  • Informed Consent Form (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/03/NCT04941703/ICF_000.pdf